CLINICAL TRIAL: NCT04153812
Title: Clinical Study on the Safety and Effectiveness of Vagus Nerve Stimulation in the Treatment of Refractory Depression
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VNS20190620
Record Dates: First submitted 2019-11-03; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Refractory Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: vagus nerve stimulation — Vagus nerve stimulation (VNS) is a new technique for stimulating the left cervical vagus nerve through implanted lead and a programmable pulse generator.

SUMMARY:
Based on the mechanism hypothesis and clinical efficacy of VNS in treating refractory depression, this study will evaluate the safety and efficacy of VNS in treating refractory depression through a small sample of clinical trials

DETAILED DESCRIPTION:
This clinical trial is a prospective, self - controlled clinical validation study. Subjects who met the inclusion criteria and did not meet the exclusion criteria were screened to enter the test. After admission, subjects received vagus nerve stimulation and conventional treatment. Enrolled 10 subjects. Parameter setting and observation were performed 2 weeks after implantation of the vagus nerve stimulation lead and pulse generator, and follow-up evaluation was performed at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. patients with treatment-resistant depression (patients with Hamilton depression scale (HAMD) score reduction rate still less than 50% after adequate treatment with two or more antidepressants)
2. age 18-65; Male or female
3. the patient has a depressive course of 2 years or more or has 2 or more major depressive episodes
4. HAMD-17 score> 17 was at baseline

Exclusion Criteria:

1. pregnant or lactating women, women of childbearing age who plan or have no safe contraceptive measures
2. a patient who is or has been diagnosed with a mental disorder other than depression; Depressive episode with psychotic symptoms
3. patients currently at serious risk of suicide
4. prior 12 months of alcohol or substance dependence, or prior 6 months of substance abuse other than nicotine
5. patients with cardiovascular diseases (myocardial infarction or cardiac arrest) and organic brain diseases (such as cerebral hemorrhage, massive cerebral infarction, encephalitis and epilepsy)
6. accept other clinical trials
7. patients requiring systemic mri after implantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
HAMD-17 | 6 months
  HAMD-17 score reduction rate at 6 months of follow-up compared to baseline

SECONDARY OUTCOMES:
HAMD-17 | 12months
  HAMD-17 score reduction rate at 3，12 months of follow-up compared to baseline
MADRS | 12months
  Changes in MADRS scores at 3, 6, and 12 months of follow-up compared to baseline
IDS-SR | 12months
  Changes in IDS-SR scores at 3, 6, and 12 months of follow-up compared to baseline
CGI | 12months
  Changes in CGI scores at 3, 6, and 12 months of follow-up compared to baseline
PSQI | 12months
  Changes in PSQI scores at 3, 6, and 12 months of follow-up compared to baseline

OTHER OUTCOMES:
safety | 12months
  The incidence of adverse events and serious adverse events at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xian, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided